CLINICAL TRIAL: NCT06734637
Title: A Single-arm, Single-center Study to Explore the Safety and Efficacy of Pegylated Interferon Alpha in Chinese Patients With ET (Essential Thrombocythemia) and PV (Polycythemia Vera).
Brief Title: Efficacy and Safety of Peginterferon in ET and PV.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhenya Hong (Other)
Responsible Party: Sponsor-Investigator, Zhenya Hong, Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024S005
Record Dates: First submitted 2024-12-11; First posted 2024-12-16 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Essential Thrombocythemia; Polycythemia Vera
Keywords: Essential thrombocythemia; Polycythemia vera; Peginterferon α-2b
MeSH Terms: conditions — Thrombocythemia, Essential; Polycythemia Vera

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Peginterferon α-2b (Experimental)
  Interventions: Drug: Peginterferon α-2b injection

INTERVENTIONS:
Drug: Peginterferon α-2b injection — Participants will receive Peginterferon α-2b 180 mcg once a week and follow-up. Dose adjustments will be made by the investigator based on the type and severity of adverse event (AE).

SUMMARY:
This is a single-arm, single-center study aims to recruit 40 participants with Essential Thrombocythemia (ET) and Polycythemia Vera (PV). Eligible participants will receive a subcutaneous injection of Peginterferon α-2b 180 mcg once a week and follow-up，and efficacy and safety will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Meet the 2016 WHO diagnostic criteria for ET (Essential Thrombocythemia) and PV (Polycythemia Vera)

   * ET (Essential Thrombocythemia) major criteria:

     1. Platelet count > 450 * 10^9/L; (2) Bone marrow biopsy shows marked megakaryocytic proliferation with increased mature megakaryocyte volume and increased nuclear lobulation. There is no significant granulocytic proliferation, left shift, or erythroid proliferation, with grade 1 fibrosis observed in a few cases; (3) Does not meet the WHO diagnostic criteria for BCR-ABL1+ CML, PV, PMF, MDS, or other myeloproliferative neoplasms; (4) JAK2, CALR, or MPL mutation positive.

        Secondary criteria: (1) Presence of a clonal marker or absence of evidence for reactive thrombocytosis.

        The diagnosis of ET requires the fulfillment of all four main criteria, or the first three main criteria plus one secondary criterion.
   * PV (Polycythemia Vera) main criteria: (1) Hemoglobin > 16.5 g/dL in males, > 16 g/dL in females, or Hematocrit > 49% in males, > 48% in females, or an increase in red cell volume of 25% or more above the normal value; (2) Bone marrow biopsy shows increased cellularity inappropriate for age, with marked erythroid, granulocytic, and megakaryocytic proliferation, and the presence of mature megakaryocytes of varying sizes and morphologies; (3) JAK2 V617F mutation positive or JAK2 exon 12 mutation positive.

   Secondary criteria: Serum Epo (Erythropoietin) level below the lower limit of the normal range.

   The diagnosis of PV requires the fulfillment of three major criteria, or the first two main criteria plus one secondary criterion.
2. For ET patients, the criteria for cytoreductive therapy must be met, as follows:

(1) For patients without a history of thrombosis: Age ≥ 60 years, regardless of the presence of cardiovascular risk (CVR) or JAK2V617 mutation; Any age with a platelet count > 1500 × 109/L. (2) For patients with a history of arterial thrombosis: Any age, regardless of the presence of CVR and JAK2V617 mutation; (3) For patients with a history of venous thrombosis: Any age, regardless of the presence of CVR and JAK2V617 mutation; 3.ECOG score ≤ 2. 4.Cardiac ejection fraction (EF) ≥ 60%. 5.The participant voluntarily signs the informed consent form.

Exclusion Criteria:

* Previous treatment with Peginterferon α-2b.
* ET patients who do not meet the criteria for cytoreductive therapy as per the 2016 Chinese Expert Consensus on Primary Thrombocythemia.
* Allergy to the active ingredient, α-interferon, or any excipients of this product.
* History of psychiatric illness, or allergy to interferon.
* Plasma total bilirubin greater than twice the normal value.
* Severe cardiac disease, liver insufficiency, chronic kidney disease, and neurological disorders (such as depression or mania).
* History of other malignant tumors within the past three years.
* Autoimmune chronic hepatitis.
* Any condition deemed unsuitable for inclusion by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-11-20 (Actual); Primary Completion 2026-11-20 (Estimated); Study Completion 2027-11-20 (Estimated)

PRIMARY OUTCOMES:
Hematologic remission rate | Week 12,24

SECONDARY OUTCOMES:
Molecular remission rate | Week 24,48
Peripheral blood driver genes | Week 24,48
Bone marrow-driven genes | Week 24,48
The incidence of thrombosis | Week 24,48
Incidence of bleeding events | Week 24,48
The incidence of progression to myelofibrosis. | Week 24,48
The incidence of acute leukemia. | Week 24,48
Changes in the burden of driver gene mutations during maintenance therapy. | Week 24,48
Hematologic remission | Week 48
Spleen enlargement remission rate. | Week 24,48

CONTACTS AND LOCATIONS:
Overall Officials: ZhenYa Hong, Ph.D, Principal Investigator — Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No